CLINICAL TRIAL: NCT00301093
Title: Vaccination for CML Patients With Persistent Disease on Imatinib Mesylate
Brief Title: Vaccine Therapy and Imatinib Mesylate in Treating Patients With Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Martha Wadleigh, M.D., Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-126; R21CA115043 (NIH); P30CA006516 (NIH); CDR0000456445 (Registry Identifier: NCI PDQ); NCT00215475 (obsolete NCT alias)
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: GM-K562 cell vaccine — Once weekly for 3 vaccination, then every other week for 3 vaccinations, and then every month for 3 vaccinations until the participant has received a total of 9 vaccinations
Drug: imatinib mesylate — Participants will continue on current dose

SUMMARY:
RATIONALE: Vaccines made from gene-modified cancer cells may help the body build an effective immune response to kill cancer cells. Imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving vaccine therapy together with imatinib mesylate may be an effective treatment for chronic myelogenous leukemia.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy when given together with imatinib mesylate in treating patients with chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of GM-K562 cell vaccine when administered with imatinib mesylate in patients with persistent chronic phase chronic myelogenous leukemia in first hematologic response.
* Determine the safety and toxic effects of GM-K562 cell vaccination in these patients.

Secondary

* Determine the disease response by serial BCR-ABL quantitative polymerase chain reaction measurements in patients treated with this regimen.
* Determine the development of tumor immunity in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of GM-K562.

Patients continue to receive oral imatinib mesylate at the same stable dose as before study entry. Patients receive GM-K562 subcutaneously on days 1, 8, 15, 29, 43, 57, 85, 113, and 141 in the absence of disease progression or unacceptable toxicity.

Cohorts of 10 patients receive escalating doses of GM-K562 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 10 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed periodically for 20 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myelogenous leukemia

  * Chronic phase disease
  * Philadelphia chromosome positive disease
* Disease in first complete hematologic response, defined by all of the following:

  * Complete normalization of peripheral blood counts with WBC < 10,000/mm^3
  * Platelet count < 450,000/mm^3
  * No immature cells (e.g., myelocytes, metamyelocytes, or blasts) in the peripheral blood
* Persistent molecular evidence of disease

  * Detectable BCR-ABL transcript by quantitative polymerase chain reaction
  * Less than 2 log reduction in peripheral blood or bone marrow BCR-ABL transcripts levels compared to a standardized baseline
* Must have received imatinib mesylate for > 1 year of which the last 3 months were at stable dose ≥ 300 mg/day

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test
* No known HIV
* ALT or AST ≤ 3 times upper limit of normal
* Oxygen saturation ≥ 93% at room air
* No history of recent acute myocardial infarction
* No history of unstable angina
* No pulmonary decomposition requiring hospitalization within the past 3 months
* No concurrent and/or uncontrolled psychiatric or medical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior allogeneic stem cell transplantation
* At least 2 months since other prior experimental therapy
* At least 6 months since prior participation in another vaccine study
* No concurrent systemic immunosuppressive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-09; Primary Completion 2007-05 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Safety and Toxicity | 3 years
  To assess the safety and toxicity of GM-K462 vaccination in CP CML patients who have acheived a complete hematologic response to imatinib.

SECONDARY OUTCOMES:
Disease Response | 3 years
  To assess disease response after GM-K562 vaccination by serial BCR-ABL Q-PCR measurements
Tumor immunity | 3 years
  To characterize the development of tumor immunity in response to vaccination with GM-K562 cells

CONTACTS AND LOCATIONS:
Overall Officials: Martha Wadleigh, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States